CLINICAL TRIAL: NCT02449161
Title: The Effect of Post Ablation Medroxyprogesterone Acetate on Endometrial Amenorrhea Rates: a RCT
Brief Title: The Effect of Post Ablation Medroxyprogesterone Acetate on Endometrial Amenorrhea Rates
Acronym: MPA postAE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Missing fund to continue
Sponsor: Guy Waddell (Other)
Collaborators: CSSS Chicoutimi (Unknown)
Responsible Party: Sponsor-Investigator, Guy Waddell, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-31-2015-998
Record Dates: First submitted 2015-05-13; First posted 2015-05-20 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Menorrhagia
Keywords: endometrial ablation
MeSH Terms: conditions — Menorrhagia | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- MPA (Experimental): medroxyprogesterone acetate, 10 mg/day, for 90 days, following endometrial ablation
  Interventions: Drug: MPA
- placebo (Placebo Comparator): 1 placebo/day, for 90 days, following endometrial ablation
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MPA
  Other Names: provera
  Arms: MPA
Drug: placebo
  Arms: placebo

SUMMARY:
Heavy menstrual bleeding are a common reason for consultation in gynecology and are defined by International Federation of Gynecology and Obstetrics as the perception of menstrual volume increased regardless of the frequency, duration and regularity. Some studies report that up to 30% of women will suffer from heavy periods during their lifetime. The first line treatment of heavy bleeding is medical. However, a significant proportion of women require surgery. Until the 80s, hysterectomy was one of the only surgical options and often performed as the first line treatment. Since twenty years now the endometrial ablation has become a preferred option for dysfunctional uterine bleeding and avoids hysterectomy in a significant proportion of patients suffering from this type of problem. Endometrial ablation is much less invasive and morbid than hysterectomy, however, many patients do not achieve a complete amenorrhea with endometrial ablation and about 15% may have to require a new intervention, such as hysterectomy, following the persistence of menstrual problems. A Cochrane review published in 2013 showed that the satisfaction rate following endometrial ablation is high at 70-80% and about 35% of women have amenorrhea. The complete destruction of the endometrium is the most important predictor of the success of the procedure. Studies have shown that better results are obtained when the surgery is performed when the endometrium is thin or immediately following menses or following administration of a hormonal agent causes atrophy of the endometrium. One of the agents studied to prepare the endometrium before ablation is medroxyprogesterone acetate (MPA) as injectables (DMPA) and oral. Progestins have an antiproliferative effect on the endometrium. In recent years, numerous studies have examined the use of various agents preoperatively, including MPA and DMPA to facilitate surgery by reducing the thickness of the endometrium. However, few studies have focused on the conditions of the post-operative period to promote the therapeutic response to the intervention. The investigators hypothesis is whether the MPA administered in immediate post-operative would inhibit proliferation of endometrial cells responsible for the persistence of menstruation and optimize the clinical response to endometrial ablation.

ELIGIBILITY:
Inclusion Criteria:

* endometrial ablation planned for eavy menstrual bleeding
* No abnormalities at hysteroscopy
* No evidence of hyperplasia or neoplasia in endometrial biopsy
* Hysterometry of ≤ 10 cm preoperatively

Exclusion Criteria:

* Any indication against MPA
* Intrauterine pathology causing heavy bleeding
* hormonal treatment provided during the postoperative period (during the first 4 months)
* preoperative hormonal therapy with a residual postoperative effect
* breastfeeding
* future pregnancy planned
* menopausal women
* endometrial ablation antecedent
* Suspected pelvic infection
* known Hematologic Disease
* Taking anticoagulant
* Taking progestin in the 6 months before surgery

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
quantification of amenorrhea | 12 months
  using the "Pictorial Blood Loss Assessment Chart" for quantification

SECONDARY OUTCOMES:
quantification of amenorrhea | 4 months
  using the "Pictorial Blood Loss Assessment Chart" for quantification
documentation of side effects | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada